CLINICAL TRIAL: NCT03618420
Title: CASPER Study: Copeptin in Adolescent Participants With Type 1 Diabetes and Early Renal Hemodynamic Function
Brief Title: Copeptin in Adolescent Participants With Type 1 Diabetes and Early Renal Hemodynamic Function
Acronym: CASPER
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-0820
Record Dates: First submitted 2018-08-01; First posted 2018-08-07 (Actual); Results first posted 2021-08-31 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-03

CONDITIONS: Diabetes Mellitus, Type 1; Nephropathy; Diabetic Nephropathies; Juvenile Diabetes; Diabetes Mellitus Complication; Autoimmune Diabetes; Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Kidney Diseases; Diabetic Nephropathies; Diabetes Complications | interventions — p-Aminohippuric Acid; Iohexol

STUDY DESIGN:
Intervention Model Description: All study participants will receive the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Clinical Investigation (Other): All participants will undergo assessment of Glomerular Filtration Rate, (Iohexol Inj 300 mg/mL) and Effective Renal Plasma Flow (Aminohippurate Sodium Inj 20%). In addition, participants will undergo imaging assessment that includes Dual X-Ray Absorptiometry (DXA), renal Blood Oxygen Level Dependent (BOLD) and Arterial Spin Labeling (ASL) MRI.
  Interventions: Drug: Aminohippurate Sodium Inj 20%; Drug: Iohexol Inj 300 mg/mL

INTERVENTIONS:
Drug: Aminohippurate Sodium Inj 20% — Diagnostic aid/agent used to measure effective renal plasma flow (ERPF)
  Other Names: Aminohippuric acid; Para-aminohippurate (PAH); Sodium 4-amino hippurate (PAH) inj 20% 2g/10 mL
Drug: Iohexol Inj 300 mg/mL — Diagnostic aid/agent used to measure glomerular filtration rate (GFR)
  Other Names: omnipaque 300

SUMMARY:
Over 1.25 million Americans have type 1 diabetes (T1D), increasing risk for early death from cardiorenal disease. The strongest risk factor for cardiovascular disease (CVD) and mortality in T1D is diabetic kidney disease (DKD). Current treatments, such as control of hyperglycemia and hypertension, are beneficial, but only partially protect against DKD.

Hyperfiltration is common in youth with T1D, and predicts progressive DKD. Hyperfiltration is also associated with early changes in intrarenal hemodynamic function, including increased renal plasma flow (RPF) and glomerular pressure. Intrarenal hemodynamic function is strongly influenced by the renin-angiotensin-aldosterone system (RAAS), which is also considered a key player in the pathogenesis of DKD. Preliminary data demonstrate differences in intrarenal hemodynamic function and RAAS activation in early and advanced DKD in T1D. However, the pathophysiology contributing to the differences observed in RAAS activation and intrarenal hemodynamic function in T1D are poorly defined Animal research demonstrates that arginine vasopressin (AVP) acts directly to modify intrarenal hemodynamic function, but also indirectly by activating RAAS. Preliminary data suggest that elevated copeptin, a marker of AVP, which predicts DKD in T1D adults, independently of other risk factors. However, no human studies to date have examined how copeptin relates to intrarenal hemodynamic function in early DKD in T1D. A better understanding of this relationship is critical to inform development of new therapies targeting the AVP system in T1D. Accordingly, in this study, the investigators propose to define the relationship between copeptin and intrarenal hemodynamics in early stages of DKD, by studying copeptin levels, renal plasma flow, and glomerular filtration in youth (n=50) aged 12-21 y with T1D duration < 10 y.

ELIGIBILITY:
Inclusion Criteria:

* Antibody+ T1D with <10 yr duration
* Age 12-21 years
* BMI ≥ 5%ile
* Weight<350 lbs and > 57 lbs.
* No anemia
* HbA1c <12%

Exclusion Criteria:

* Severe illness, recent diabetic ketoacidosis (DKA)
* Estimated Glomerular Filtration Rate (eGFR) <60ml/min/1.73m2 or creatinine > 1.5mg/dl or history of ACR≥300mg/g
* Anemia or allergy to shellfish or iodine
* Pregnancy or nursing
* MRI scanning contraindications (claustrophobia, implantable devices, >350 lbs)
* Angiotensin-converting enzyme (ACE) inhibitors, angiotensin receptor blockers (ARB), diuretics, sodium-glucose co-transport (SGLT) 2 or 1 blockers, daily NSAIDs or aspirin, sulfonamides, procaine, thiazolsulfone or probenecid, atypical antipsychotics and steroids

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-10-19 (Actual); Study Completion 2021-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Petter Bjornstad, MD, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pauley ME, Vinovskis C, MacDonald A, Baca M, Pyle L, Wadwa RP, Fornoni A, Nadeau KJ, Pavkov M, Nelson RG, Gordin D, de Boer IH, Tommerdahl KL, Bjornstad P. Triglyceride content of lipoprotein subclasses and kidney hemodynamic function and injury in adolescents with type 1 diabetes. J Diabetes Complications. 2023 Feb;37(2):108384. doi: 10.1016/j.jdiacomp.2022.108384. Epub 2022 Dec 13. PMID 36623423
- [Derived] Vigers T, Vinovskis C, Li LP, Prasad P, Heerspink H, D'Alessandro A, Reisz JA, Piani F, Cherney DZ, van Raalte DH, Nadeau KJ, Pavkov ME, Nelson RG, Pyle L, Bjornstad P. Plasma levels of carboxylic acids are markers of early kidney dysfunction in young people with type 1 diabetes. Pediatr Nephrol. 2023 Jan;38(1):193-202. doi: 10.1007/s00467-022-05531-3. Epub 2022 May 4. PMID 35507146
- [Derived] Vinovskis C, Li LP, Prasad P, Tommerdahl K, Pyle L, Nelson RG, Pavkov ME, van Raalte D, Rewers M, Pragnell M, Mahmud FH, Cherney DZ, Johnson RJ, Nadeau KJ, Bjornstad P. Relative Hypoxia and Early Diabetic Kidney Disease in Type 1 Diabetes. Diabetes. 2020 Dec;69(12):2700-2708. doi: 10.2337/db20-0457. Epub 2020 Jul 31. PMID 32737116

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clinical Investigation
Started (Study Start and IRB Approval) | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Clinical Investigation
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.0 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black non-Hispanic | 1
  Hispanic | 3
  White non-Hispanic | 46

OUTCOME MEASURES:

1. Primary Outcome: Copeptin Levels
Description: Measured by fasting blood draw; Copeptin will be measured by ultrasensitive assays on KRYPTOR Compact Plus analyzers using the commercial sandwich immunoluminometric assays (Thermo Fisher Scientific, Waltham, MA). The copeptin assay has a lower limit of detection of 0.9 pmol/L, and a sensitivity of <2pmol/L. Elevated copeptin will be defined as >13pmol/L, which is >97.5th percentile for healthy adults (68).
Time Frame: 4 hours
Population: The overall number of participants analyzed for the outcome measure Copeptin levels is 49 because of an assay issue, specifically one of the samples failed during quality control.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Clinical Investigation
Number analyzed (Participants) | 49
pmol/L | 8.3 (5.0)

2. Primary Outcome: Effective Renal Plasma Flow (ERPF)
Description: Measured by para-aminohippurate (PAH) clearance; An intravenous (IV) line was placed, and participants were asked to empty their bladders. Spot plasma and urine samples were collected prior PAH infusion. PAH (2 g/10 mL, prepared at the University of Minnesota, with a dose of [weight in kg]/75 × 4.2 mL; IND #140129) was given slowly over 5 min followed by a continuous infusion of 8 mL of PAH and 42 mL of normal saline at a rate of 24 mL/h for 2 h. After an equilibration period, blood was drawn at 90 and 120 min, and ERPF was calculated as PAH clearance divided by the estimated extraction ratio of PAH, which varies by the level of GFR (13). We report absolute ERPF (mL/min) in the main analyses because the practice of indexing ERPF for body surface underestimates hyperperfusion, and body surface area (BSA) calculations introduce noise into the clearance measurements.
Time Frame: 4 hours
Population: The overall number of participants analyzed for the outcome measure ERPF is 37 because PAH was unavailable for several of the first study visits.
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Clinical Investigation
Number analyzed (Participants) | 37
ml/min | 820 (125)

3. Primary Outcome: Glomerular Filtration Rate (GFR)
Description: Measured by iohexol clearance; An intravenous (IV) line was placed, and participants were asked to empty their bladders. Spot plasma and urine samples were collected prior to iohexol infusion. Iohexol was administered through bolus IV injection (5 mL of 300 mg/mL; Omnipaque 300, GE Healthcare). An equilibration period of 120 min was used and blood collections for iohexol plasma disappearance were drawn at +120, +150, +180, +210, +240 min (11). Because the Brøchner-Mortensen equation underestimates high values of GFR, the Jødal-Brøchner-Mortensen equation was used to calculate the GFR (12). We report absolute GFR (mL/min) in the main analyses because the practice of indexing GFR for body surface underestimates hyperfiltration, and body surface area (BSA) calculations introduce noise into the clearance measurements.
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Clinical Investigation
Number analyzed (Participants) | 50
ml/min | 189 (40)

4. Secondary Outcome: Renal Perfusion
Description: Measured by Arterial Spin Labeling (ASL) MRI; ASL MRI: ROI analysis will be used to estimate (delta) M (difference in signal intensity between non-selective and selective inversion images). Using the same ROI, M0 will be estimated from the proton density image. T1 measurements from the same ROI will be obtained by fitting the signal intensity vs. inversion time data as described previously (104) using XLFit (ID Business Solutions Ltd., UK) or T1 maps created using MRI Mapper (Beth Israel Deaconess Medical Center, Boston). Partition coefficient will be assumed to be 0.8 ml/gm (105, 106). These values will then be used to estimate regional blood flow.
Time Frame: 10 min
Population: The overall number of participants analyzed for the outcome measure Renal Perfusion is 45 because scans did not meet the high quality control standard of our MRI reader and thus were omitted.
Measure: Mean (Standard Deviation); unit: ml/min/100g
Arm/Group | Clinical Investigation
Number analyzed (Participants) | 45
ml/min/100g | 180 (39)

5. Secondary Outcome: Renal Oxygenation
Description: Measured by Blood Oxygen Level Dependent (BOLD) MRI; Regions of interest (ROI) analysis for BOLD MRI will be performed on a Leonardo Workstation (Siemens Medical Systems, Germany). Typically, 1 to 3 regions in each, cortex and medulla, per kidney per slice will be defined leading to a total of about 10 ROIs per region (cortex and medulla) per subject. The mean and standard deviation of these 10 measurements will be used a R2* measurement for the region, for the subject and for that time point. These data are used to calculate kidney oxygen availability (R2*), which is the BOLD-MRI outcome.
Time Frame: 60 min
Population: The overall number of participants analyzed for the outcome measure Renal Oxygenation is 41 because scans did not meet the high quality control standard of our MRI reader and thus were omitted.
Measure: Mean (Standard Deviation); unit: s^-1
Arm/Group | Clinical Investigation
Number analyzed (Participants) | 41
s^-1 | 22.7 (2.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 1 month post procedure (since this was a cross-sectional study).
Arm/Group | Clinical Investigation
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 2/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clinical Investigation (N=50)
Vasovagal syncope (Vascular disorders) | 1 — Participant experienced vasovagal syncope as a result of anxiety and peripheral intravenous line (PIV) placement at the beginning of study visit; known risk which is included in the consent form.
Headache/lightheadedness/nausea (Nervous system disorders) | 1 — Participant experienced headache and lightheadedness during screening visit when blood draw to obtain screening labs was attempted. This is a known risk which is included in the consent form.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT03618420/Prot_SAP_000.pdf